CLINICAL TRIAL: NCT01220505
Title: A Post Market Surveillance Validation to Evaluate the Effectiveness of the Following System: Polaris Deformity Spinal System
Brief Title: Post Market Surveillance to Evaluate the Effectiveness the Polaris Deformity Spinal System
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-058
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Spinal Deformity
Keywords: scoliosis; kyphosis; spinal deformity; curvature; lordosis
MeSH Terms: conditions — Scoliosis; Kyphosis; Lordosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Surgery — All subjects will have spinal surgery between the levels of T1 and Ilium using the Polaris Deformity Spinal System
  Other Names: Polaris Deformity Spinal System; Trivium Deformtiy Correction System

SUMMARY:
The purpose of this Post Market Surveillance Validation is to document the performance and clinical outcomes of the Polaris Deformity Spinal System & Trivium 3D Spinal Deformity Correction System.

DETAILED DESCRIPTION:
The purpose of this Post Market Surveillance Validation is to document the performance and clinical outcomes of the Polaris Deformity Spinal System & Trivium 3D Spinal Deformity Correction System. We have extended the study tol collect further outcomes data at the 12 month time point.

ELIGIBILITY:
Inclusion Criteria:

* 200 subjects at 10 clinical centers.
* All subjects undergoing spinal fusion surgery between the levels of T1- Ilium (Thoracic 1 to Ilium)
* All subjects are skeletally mature with spinal deformity.
* Risser score must be ≥ 3.
* Subjects or their representative must be willing and able to give informed consent and assent (if applicable).
* Subjects who do not meet any of the following contraindications: spinal infection or inflammation, morbid obesity, mental illness, alcoholism, drug abuse, pregnancy, metal sensitivity, foreign body sensitivity, patients with inadequate tissue coverage over the operative site, open wounds local to the operative area, any case not described in the specific indications

Exclusion Criteria:

* Any subject who does not meet the inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with a spinal defomrity with a Risser score of a minimum of 3 where the physician has determined that the patient requires a spinal fusion of the thoracic or lumbar spine are eligible for entry into the post market surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Maintenance of Deformity Correction | 6 months
  The primary outcome measure for this trial will be the percentage of subjects who have maintained their degree of deformity correction within 10% from immediate post-op to the 6 month follow-up visit.

SECONDARY OUTCOMES:
Decreased Operative Time | 6 Months
  Comparison of Operative times vs. literature

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Stinson, Study Director — Zimmer Biomet
Locations (6):
- United States (5):
  - Orthopedics for Kids, PC, Birmingham, Alabama
  - Loma Linda University, Loma Linda, California
  - Children's Orthopedics of Atlanta, Atlanta, Georgia
  - Orthopedics Indianapolis, P.C., Indianapolis, Indiana
  - Rochester Hills Orthopedics, Rochester Hills, Michigan
- Torre Auxillo Mutuo, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Undecided